CLINICAL TRIAL: NCT07123831
Title: The Effect of Privacy Education With Virtual Reality Application on Children's Privacy Awareness and Saying No Skills
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yuzuncu Yil University (Other)
Responsible Party: Principal Investigator, Ayşe Deniz, Hemşire, Yuzuncu Yil University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2024\07-39
Record Dates: First submitted 2025-07-19; First posted 2025-08-14 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Privacy Education
Keywords: Children, Privacy, Saying No, Privacy Education, VR

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- No Intervention Group (No Intervention): no intervention in the control group
- VR-Based Privacy Education (Experimental): the experimental group was provided with virtual reality glasses supported privacy training
  Interventions: Other: virtual reality supported privacy education

INTERVENTIONS:
Other: virtual reality supported privacy education — The experimental group was shown a video with virtual reality application for 15 minutes in an empty classroom environment determined in the primary school at a time and in a way that would not disrupt the lessons. Then, verbal expression, question-answer and feedback were given for 10 minutes. After this training session, the experimental group was repeated twice with virtual reality goggles at two-week intervals and their questions were answered. No intervention was made to the students in the control group. At the end of the sixth week, the researcher administered post-tests to each student in the experimental and control groups.
  Arms: VR-Based Privacy Education

SUMMARY:
This study was conducted to evaluate the effect of virtual reality (VR)-based privacy education on 4th grade students' privacy awareness (PA) and ability to say no (SN) levels. The study was conducted in a primary school affiliated to the Ministry of National Education in a province in the Eastern Anatolia Region between November 2024 and May 2025 with a pretest/posttest control group. The population of the study consists of 4th grade students studying in primary schools in the province. The school where the data were collected was determined by lottery method among the schools that met the sample size.In the G*Power analysis, it was calculated that 88 students would be sufficient, but the study was completed by including 97 students. The experimental (S=46) and control groups (S=51) were determined by lottery. Students in the experimental group were given privacy training using Peeq SC-AI05 virtual reality (VR) goggles. Child Descriptive Information Form, Privacy Awareness Scale for Primary School Students (PAS) and Ability to Say No Scale for Children (NS) were used as data collection tools.Data were analyzed with SPSS V26 program. Ethical principles were adhered to during the research process.

ELIGIBILITY:
Inclusion Criteria:The student verbally expresses his/her willingness to participate,

* Parent's approval of the informed consent form,
* Being in the fourth grade at primary school level,
* The inclusion criteria were that the student was open to communication and did not have any psychological or chronic health problems.

Exclusion Criteria:Those who do not want to participate in the research and those who want to withdraw during the research process

- Incomplete completion of the scale or questionnaire

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 97 (Actual)
Dates: Start 2024-11-19 (Actual); Primary Completion 2025-03-31 (Actual); Study Completion 2025-05-30 (Actual)

PRIMARY OUTCOMES:
Privacy Consciousness Scale for Elementary School Students | 20weeks
  The scale consists of 16 items and 4 factors. These factors are named as "Personal Security ", "Sharing Personal Information", "Social Media Privacy" and "Parental Control". Students were asked to answer the statements in the items with a 3-point Likert scale as "disagree", 'undecided' and "agree". The scale will be scored as 1 point for each disagree response, 2 points for an undecided response and 3 points for an agree response. The score that can be obtained from the scale varies between 16 and 48 points. Higher scores indicate higher privacy awareness. There are 2 reverse items in the scale. The Cronbach's alpha internal consistency coefficient of the Privacy Consciousness Scale for Elementary School Students was reported to be .86.

SECONDARY OUTCOMES:
The Ability to Say "No" Scale for Children | 20weeks
  The scale aims to measure the ability of 4th grade primary school students to say "no". This scale consists of the refusal subscale and the resistance subscale. The refusal and resistance sub-dimensions of the scale consist of 6 items each. refusal subscale includes items to measure whether students can say "no" in the face of demands, reactions and behaviors that they do not like or find unreliable. On the other hand, the resistance subscale includes items to determine whether students step back in the face of the motivational efforts they may encounter with the emotions they experience after saying "no". The students were asked to answer the statements contained in the items on a 5-point Likert scale as "never", "rarely", 'sometimes', "most of the time" and "always". In the evaluation of the scores obtained from the SN, the coding for the refusal dimension is scored as it is, while the coding for the resistance dimension is scored in reverse.

CONTACTS AND LOCATIONS:
Locations (1):
- A primary school affiliated to the Ministry of National Education in Van province, Van, Tuşba, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes